CLINICAL TRIAL: NCT05375019
Title: The Effectiveness of a Positive Discipline Program Applied To The Parents of Preschool Children: A Randomized Controlled Study
Brief Title: Positive Discipline in Parent Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Hatice Dayilar Candan, principal investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ege HDCandan
Record Dates: First submitted 2022-05-03; First posted 2022-05-16 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Parenting
Keywords: Positive discipline; preschool period; parent training; parenting attitudes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (positive discipline program) (Experimental): The intervention group was provided with 8 weekly sessions of a 90 minutes positive discipline program.
  Interventions: Behavioral: Positive discipline program
- Active control group (free interaction) (Active Comparator): while the active control group was provided with 8 weekly 90 minute sessions of free interaction.
  Interventions: Behavioral: active control group
- No-contact group (No Intervention): No intervention was performed with the no-contact control group.

INTERVENTIONS:
Behavioral: Positive discipline program — The intervention group was provided with 8 weekly sessions of a 90 minutes positive discipline program
  Arms: Intervention group (positive discipline program)
Behavioral: active control group — free interaction group consisting of topics determined by the families.
  Arms: Active control group (free interaction)

SUMMARY:
The aim of this study was to examine the effectiveness of a Positive Discipline Program applied to the parents of preschool children. Accordingly, the tertiary aims of this study included determining the effects of a positive discipline program on the child upbringing attitudes of parents with preschool children, their perceptions regarding each other's child upbringing attitudes, and the communication between preschool children and their parents.

DETAILED DESCRIPTION:
This randomized controlled experimental study included pretest, posttest, and monitoring test applications with an intervention group, an active control group, and a no-contact control group. The study was conducted between May 2020 and June 2022. The universe of the study consisted of 653 parents with preschool (ages 3-6) children registered to the Izmir Bornova Şükrü Ergil Family Health Center No:9. Sample size was calculated using power analysis and assigned randomly to the intervention, active control, and no-contact control groups in groups of 24 (n=72). The intervention group was provided with 8 weekly sessions of a 90 minutes positive discipline program while the active control group was provided with 8 weekly 90 minute sessions of free interaction. No intervention was performed with the no-contact control group. Data collection was performed using a Personal Information Form, Parental Attitude Scale (PAS), Assessment of Parenting Attitudes of Couples Scale (APACS) and the Parent Child Communication Scale (PCCS).

ELIGIBILITY:
Inclusion Criteria:

* Registered at Şükrü Ergil Family Health Center No. 9 in Bornova,
* Agreeing to participate in the research,
* Having children between the ages of 3-6,
* Parents have not participated in any parent education program before,
* Having the cognitive ability to receive education,
* Able to read and write,
* Having no problems in hearing, seeing and understanding,
* Will be able to participate in at least 7 sessions of the positive discipline program and active control group,
* Capable of using an online program (because it is made online).

Exclusion Criteria:

* Failure to attend at most one of the positive training program and active control group sessions,
* Parent's request to withdraw at any stage of the trial.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
improvement in parenting attitudes | 8 weeks later
  Parental Attitude Scale (PAS) was used that scale consists of three sub-dimension. The 38-item scale has three sub-dimensions: "13 items Democratic Attitude", "10 items Oppressive and Authoritarian Attitude", and "12 items Overprotective Attitude". A high score in each dimension means that the attitude characteristic related to that sub-dimension is dominant. It is expected that this study will change in oppressive and authoritarian, overprotective and democratic parenting attitude.
improvement in Parenting Attitudes of Couples | 8 weeks later
  Assessment of Parenting Attitudes of Couples Scale (APACS) was used that scale consist of four sub-dimension. The scale, which consists of 50 items in total, has four sub-dimensions: "15 items Democratic Attitude", "14 items Oppressive and Authoritarian Attitude", "10 items Overprotective Attitude" and "11 items Permissive Attitude". Higher scores on the APACS indicate that the spouses' child rearing attitudes in the relevant sub-dimension are more dominant by observing the other parent. It is expected that this study will change in these parenting attitude.
improvement a parent's relationship with their child | 3 months later
  Parent Child Communication Scale (PCCS) was used. The parent version of the PCCS involved a 20-item measure that also consisted of a five-point scale ranging from 'almost never' to 'almost always'. This PCCS parent version is composed of four sub-scales: parent communication, parent restricted topics, child/empathy listening, and child emotional expression.I It is understood that the higher the score obtained from the scale, the higher the level of communication of the parent with his/her child. It is expected that this study will change in parent's relationship with their child.

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Eksioglu, PhD. Dr., Study Chair — TAEK
Locations (1):
- Ege University, TAEK, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
I finished my thesis and published it in Journal of Pediatric Nusing. I can share my published article.
Supporting Information: Study Protocol
Time Frame: starting starting 6 months after publication
Access Criteria: psychiatric nurse
URL: https://www.sciencedirect.com/science/article/abs/pii/S0882596323001458